CLINICAL TRIAL: NCT02026388
Title: Rare Kidney Stone Consortium Biobank, Rare Diseases Clinical Research Network
Brief Title: Rare Kidney Stone Consortium Biobank
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lieske, Principal Investigator, Mayo Clinic
Other Study IDs: 11-005413
Record Dates: First submitted 2013-12-30; First posted 2014-01-03 (Estimated); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Primary Hyperoxaluria; Dent Disease; APRT Deficiency; Cystinuria
Keywords: PH; primary hyperoxaluria; hyperoxaluria; primary oxalosis; Primary Hyperoxaluria Type 1; Primary Hyperoxaluria Type 2; Primary Hyperoxaluria Type 3; Dent; Dents; Dent Disease; Dent 1; Dent 2; Cystinuria; APRT; APRT deficiency; Biobank
MeSH Terms: conditions — Hyperoxaluria, Primary; Dent Disease; Adenine phosphoribosyltransferase deficiency; Cystinuria; Hyperoxaluria; Primary hyperoxaluria type 1; Primary hyperoxaluria type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, blood and tissue samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Primary Hyperoxaluria: Diagnosis of Primary Hyperoxaluria, or a family member of someone with this diagnosis.
- Dent Disease: Diagnosis of Dent Disease, or a family member of someone with this diagnosis.
- Cystinuria: Diagnosis of Cystinuria, or a family member of someone with this diagnosis.
- APRT deficiency: Diagnosis of APRT Deficiency, or a family member of someone with this diagnosis.

SUMMARY:
This study is being done to obtain samples from patients with primary hyperoxaluria, cystinuria, adenine phosphoribosyl transferase (APRT) deficiency, and Dent disease, and from their family members, for use in future research.

DETAILED DESCRIPTION:
Biologic samples will be stored in the biobank from well characterized patients with primary hyperoxaluria, cystinuria, APRT deficiency, and Dent disease, and from their family members, for use in future research. This will help to advance our understanding of disease expression and the factors associated with kidney injury in these four diseases with the overall goal of developing new treatments to preserve kidney function and reduce nephrocalcinosis and stone formation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary hyperoxaluria (PH) meeting one or more of the following criteria:

  1. Liver biopsy documenting alanine-glyoxylate aminotransferase (AGT) activity below the normal reference range confirming PH type 1 OR Liver biopsy documenting glyoxylate reductase/hydroxypyruvate reductase (GR/HPR) activity below the normal reference range confirming PH type 2
  2. Molecular genetic analysis (DNA testing) confirming mutations known to cause PH type 1, PH type 2, or PH type 3
  3. Urinary oxalate excretion of greater than 0.8 mmol/1.73 m2/day (>70 mg/1.73 m2/day) in the absence of a identifiable causes of secondary hyperoxaluria, including gastrointestinal disease known to cause enteric hyperoxaluria
  4. A patient in end stage kidney failure, in whom neither a liver biopsy nor mutational analysis are available must have: (a) A plasma oxalate concentration of greater than 60 umol/L and a kidney biopsy confirming extensive oxalate deposits OR (b) Evidence of systemic oxalosis
  5. Participants in the previous protocol "Tissue Bank of Urine, Blood, and Tissue Samples Collected from the Patients with Primary Hyperoxaluria" 'Mayo IRB #' #80-04. They have already consented to bank their samples and that consent will serve to enroll them in this study.
* Diagnosis of Dent disease meeting one or more of the following criteria:

  1. Identified mutation of the gene that encodes for chloride exchange transporter 5 (CLCN5)
  2. Low molecular weight proteinuria and hypercalciuria
  3. Low molecular weight proteinuria and nephrocalcinosis
* Diagnosis of APRT disease meeting one or more of the following criteria:

  1. Suspected dihydroxyadeninuria and absent APRT enzyme activity measured in red blood cells (RBCs).
  2. Homozygosity, or compound heterozygosity, for known disease-causing APRT mutations.
  3. Passage of dihydroxyadenine stones (confirmed with stone analysis).
* Diagnosis of Cystinuria meeting one or more of the following criteria:

  1. Stone analysis demonstrating that the stone contains cystine
  2. Increased urinary cystine excretion (>250 mg/gm creatinine)
* Relative of someone with confirmed primary hyperoxaluria, Dent disease, APRT deficiency (also known as dihydroxyadeninuria), or cystinuria

Exclusion Criteria:

1. Stone formers who do not meet the inclusion criteria for primary hyperoxaluria, cystinuria, Dent disease, or APRT deficiency.
2. Unwilling or unable to provide consent/assent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a confirmed Diagnosis of Primary Hyperoxaluria, Dent Disease, APRT deficiency or Cystinuria. Family members of individuals with these four diseases.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2013-05; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Number of samples stored in tissue bank | 4 years
  encourage more research

CONTACTS AND LOCATIONS:
Overall Officials: John C Lieske, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Biospecimens repository only. No individual data available to share.

REFERENCES:
- See also: Rare Kidney Stone Consortium — http://www.rarekidneystones.org/